CLINICAL TRIAL: NCT02203890
Title: Study on the Normative State and Inter- and Intra-individual Variation in Growth, Hematology, Hydration and Markers of Oxidation, Infection and Inflammation in Preschool Children With a Similar Dietary Intake
Brief Title: Normative State and Variation in Growth, Hematology, Hydration, Oxidation, Infection, Inflammation, Guatemalan Children
Status: Completed | Type: Observational
Sponsor: María José Soto (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor-Investigator, María José Soto, PhD student and nutrition researcher, Center for Studies of Sensory Impairment, Aging and Metabolism
Organization: Center for Studies of Sensory Impairment, Aging and Metabolism (Other)
Other Study IDs: CeSSIAM_02
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Growth; Hematology; Hydration; Oxidation; Infection; Inflammation; Guatemalan children
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, feces, saliva and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Apparently Healthy: Apparently healthy preschool children who attend 3 daycare centers of the Secretariat of Beneficials Works of the First Lady in Guatemalan Western Highlands

SUMMARY:
This study will provide the researchers with an opportunity for the investigation of the biomarkers and different human biology component variable interactions in children; information that can generate new correlations between markers not known at the moment.

Regarding their analysis, variation could have multiple connotations. A categorical that refers to a specific state, established with a diagnostic standard. And a numerical, referring to a range or the absolute value limits in a continuous spectrum; this research will allow us to express variability in the distance amplitude of the obtained values level, as well as classifications or categories previously established in the possible cases.

OBJECTIVES PRINCIPAL OBJECTIVE

To estimate the inter and intra-individual variety in a selected series or biological variables determinant of growth, body composition, infection, oxidation, inflammation and hydration, in preschool children sharing the same institutional-based diet.

SPECIFIC OBJECTIVES

* To determine the inter and intra-individual variation of growth in preschool children, with a similar diet, who attend Secretariat of Beneficial Works of the First Lady system daycare centers and to compare between semi-urban and rural.
* To describe the inter-individual variation of the red blood cells circulating mass in preschool children, with a similar diet, who attend day care centers and to compare between semi-urban and rural.
* To determine the inter-individual variation of systemic and intraintestinal oxidation in preschool children, with a similar diet, who attend daycare centers and to compare between semi-urban and rural.
* To describe the inter-individual variation of systemic and intraintestinal inflammation in preschool children, with a similar diet, who attend daycare centers and to compare between semi-urban and rural.
* To determine the inter and/or intra-individual variation of urinary tract infection and gastrointestinal parasite infestation in preschool children, with a similar diet, who attend daycare centers and to compare between semi-urban and rural.
* To describe the inter and intra-individual variation of the hydration status in preschool children, with a similar diet, who attend daycare centers and to compare between semi-urban and rural.
* To explore intra-individual associations in variables of the same research component or different component variables.

DETAILED DESCRIPTION:
Please note protocol is also available in Spanish.

ELIGIBILITY:
Inclusion Criteria:

* To be attending one of the SOSEP systems assigned daycare centers
* To maintain an attendance of 80% during the 8 weeks of the fieldwork
* Aged 23 to 84 months
* Being apparently healthy and with no dietary restrictions related to the foods offered with the SOSEP menu.

Exclusion Criteria:

* Children whose parents of caregivers did not sign a consent form
* Children who refused to participate in the study
* Children who refused to adhere to the collections routines.

Ages: 23 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Apparently healthy children who attend 3 daycare centers (one semi-urban, one urban-marginal and one rural) from the Secretariat of Beneficial Works of the First Lady (SOSEP) system in the Western Highlands in Quetzaltenango, Guatemala.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Weight | 7th week of observation
  Growth, measured trough weight (kg)
Hemoglobin | 8th week of observation
  Hemoglobin (mg/dl) measured in Biochemistry Laboratory in La Democracia Hospital, Quetzaltenango, Guatemala.
Urine Osmolality-1 | 6th week of observation
  Hydration Status= measured in 24-h urine through urine volume and osmolality in osmometer Model Löser 815. Results in mOsm/kg.
Height | 7th week of observation
  Growth, measured trough height (cm).
Urine Osmolality-2 | 7th week of observation
  Hydration Status= measured in 24-h urine through urine volume and osmolality Osmometer Model Löser 815. Results in mOsm/kg.
Urine Osmolality-3 | 8th week of observation
  Hydration Status= measured in 24-h urine through urine volume and osmolality in two different osmometers (Löser 815 and Osmomat 030). Results in mOsm/kg.
Urine Urea | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  urea (mg/l)
Urine Uric Acid | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  uric acid (mg/l)
Urine Sodium | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  sodium (mg/l)
Urine Potassium | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  potassium (mg/l)
Urine Calcium | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  calcium (mg/l)
Urine Magnesium | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  magnesium (mg/l)
Urine Phosphorus | 8th week of oservation
  Urine solutes measured by the Scientific Instrumentation Center from the Granada University, Spain:
  inorganic phosphorus (mg/l)
Urine 15-f2t-Isoprostanes | 8th week of observation
  Urine Oxidation biomarkers:
  15-f2t-Isoprostanes (ng/mL) Measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada using ELISA assay kit (Oxford Biomedical Research, Inc., Catalog # EA84.102606, Michigan, USA)
Urine 8-Hydroxydeoxyguanosine | 8th week of observation
  Urine Oxidation biomarkers:
  8-Hydroxydeoxyguanosine (ng/mL) Measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada using ELISA assay kits (JaICA, Nikken SEIL Co., Ltd, Catalog# IM-KOGHS 040914E, Shizouka, Japan).
Catalase Activity | 8th week of observation
  Activity of antioxidant enzymes in red blood cells; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using ELISA system:
  Catalase Activity (nmol/seg/g Hb)
Superoxide Dismutase Activity | 8th week of observation
  Activity of antioxidant enzymes in red blood cells; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using ELISA system Superoxide Dismutase Activity (U/g Hb)
Gluthathione Reductase | 8th week of observation
  Activity of antioxidant enzymes in red blood cells; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using ELISA system Gluthathione Reductase Activity (umol/min/g Hb)
Gluthathione Peroxidase | 8th week of observation
  Activity of antioxidant enzymes in red blood cells; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using ELISA system Gluthathione Peroxidase Activity (uU/g Hb)
Retinol | 8th week of observation
  Content of antioxidant compounds in plasma; Scientific Instrumentation Center, University of Granada.
  Retinol (mg/dl)
Alpha-tocopherol | 8th week of observation
  Content of antioxidant compounds in plasma; Scientific Instrumentation Center, University of Granada.
  Alpha-tocopherol (mg/l)
Beta-Carotenes | 8th week of observation
  Content of antioxidant compounds in plasma; Scientific Instrumentation Center, University of Granada.
  Beta-carotenes (mg/l)
Coenzyme Q9 | 8th week of observation
  Content of antioxidant compounds in plasma; Scientific Instrumentation Center, University of Granada.
  Coenzyme Q9 (mg/l)
Coenzyme Q10 | 8th week of observation
  Content of antioxidant compounds in plasma; Scientific Instrumentation Center, University of Granada.
  Coenzyme Q10 (mg/l)
Plasma Interleukin-1B | 8th week of observation
  Plasma Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Plasma IL-1B (pg/ml)
Plasma Interleukin-6 | 8th week of observation
  Plasma Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Plasma IL-6 (pg/ml)
Plasma Interleukin-8 | 8th week of observation
  Plasma Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Plasma IL-8 (pg/ml)
Plasma Interleukin-10 | 8th week of observation
  Plasma Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Plasma IL-10 (pg/ml)
Plasma Tumor Necrosis Factor-Alpha | 8th week of observation
  Plasma Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Plasma Tumor Necrosis Factor-Alpha (pg/ml)
Saliva Interleukin-1B | 8th week of observation
  Saliva Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system: Saliva IL-1B (pg/ml)
Saliva Interleukin-6 | 8th week of observation
  Saliva Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system: Saliva IL-6 (pg/ml)
Saliva Interleukin-8 | 8th week of observation
  Saliva Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system: Saliva IL-8 (pg/ml)
Saliva Interleukin-10 | 8th week of observation
  Saliva Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system Saliva IL-10 (pg/ml)
Saliva Tumor Necrosis Factor-Alpha | 8th week of observation
  Saliva Interleukines; measured at the Institute of Nutrition and Food Technology, Center of Biomedical Research, University of Granada, using the Luminex system:
  Saliva Tumor Necrosis Factor-Alpha (pg/ml)
Fecal Calprotectin | 8th week of observation
  Fecal Calprotectin (mg/kg) measured using the ELISA assay kit from Calpro-Lab (Catalog # CAL0100).
Intestinal Parasitosis | 8th week of observation
  Intestinal Parasitosis, measured by Biochemistry Laboratory, La Democracia Hospital, Quetzaltenango, Guatemala. Parasite cysts presence in feces.
Giardiasis Infection Presence-1 | 7th week of observation
  Analyses done by ELISA assay kit (ProSpecT Giardia EZ, catalog #R2458596), absorbance (O.D)
Giardiasis Infection Presence-2 | 8th week of observation
  Analyses done by ELISA assay kit (ProSpecT Giardia EZ, catalog #R2458596), absorbance (O.D)
White Urine Cell Count | 8th week of observation
  White urine cell count (per field), to be determined in Biochemistry Laboratory in La Democracia Hospital, Quetzaltenango Guatemala.
White Blood Cell Count | 8th week of observation
  White blood cell count (cells/ul), to be determined in Biochemistry Laboratory in La Democracia Hospital, Quetzaltenango Guatemala.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J. Soto-Méndez, MSc, Principal Investigator — Center for Studies of Sensory Impairment, Aging and Metabolism
Locations (1):
- Center for Studies of Sensory Impairment Aging and Metabolism, Guatemala, Departamento de Quetzaltenango, Guatemala

REFERENCES:
- [Result] Soto-Méndez M, Campos-Oliva R, Aguilera C, Solomons N, Schümann K, Gil A. Urinary osmolality of preschool children with a largely common weekday meal offering, from the western highlands of Guatemala. Spanish J Community Nutr. 20:13-9, 2014.
- [Derived] Soto-Mendez MJ, Romero-Abal ME, Schumann K, Gil A, Solomons NW. Normative Fecal Calprotectin Concentrations in Guatemalan Preschoolers Are High Relative to Children Reported Elsewhere. J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):238-244. doi: 10.1097/MPG.0000000000001241. PMID 27101538
- [Derived] Soto-Mendez MJ, Aguilera CM, Campana-Martin L, Martin-Laguna V, Schumann K, Solomons NW, Gil A. Variation in hydration status within the normative range is associated with urinary biomarkers of systemic oxidative stress in Guatemalan preschool children. Am J Clin Nutr. 2015 Oct;102(4):865-72. doi: 10.3945/ajcn.114.105429. Epub 2015 Aug 12. PMID 26269363
- [Derived] Soto-Mendez MJ, Aguilera CM, Mesa MD, Campana-Martin L, Martin-Laguna V, Solomons NW, Schumann K, Gil A. Interaction of Giardia intestinalis and Systemic Oxidation in Preschool Children in the Western Highlands of Guatemala. J Pediatr Gastroenterol Nutr. 2016 Jul;63(1):118-22. doi: 10.1097/MPG.0000000000000891. PMID 26111297